CLINICAL TRIAL: NCT07267026
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, First-In-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Oral Doses of SK-09 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety, Tolerability and PK of SK-09
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Consun Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PR-CR-SK(09)-101
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: FSGS; MCD
MeSH Terms: conditions — Macular dystrophy, corneal type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SK-09 (Experimental): Part 1 SAD：Six sequential dose groups will be evaluated, with the planned dose levels as follows: 20 mg, 50 mg, 100 mg, 200 mg, 400 mg, and 500 mg.
  Part 2 MAD：Three dose groups (low/medium/high, based on Part 1 SAD results) will be sequentially evaluated.
  Interventions: Drug: SK-09
- Placebo (Placebo Comparator): Part 1 SAD：Six sequential dose groups will be evaluated, with the planned dose levels as follows: 20 mg, 50 mg, 100 mg, 200 mg, 400 mg, and 500 mg.
  Part 2 MAD：Three dose groups (low/medium/high, based on Part 1 SAD results) will be sequentially evaluated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SK-09 — Dose groups of 20 mg, 50 mg, 100 mg, 200 mg, 400 mg, and 500 mg were given.
  Arms: SK-09
Drug: Placebo — Dose groups of 20 mg, 50 mg, 100 mg, 200 mg, 400 mg, and 500 mg were given.
  Arms: Placebo

SUMMARY:
This Phase 1 trial consists of two parts: Part 1 is a Single Ascending Dose (SAD) study, and Part 2 is a Multiple Ascending Dose (MAD) study. Both parts adopt a randomized, double-blind, placebo-controlled design.

DETAILED DESCRIPTION:
Part 1 is a randomized, double-blind, placebo-controlled SAD study to evaluate the safety, tolerability, PK, and PD of single oral doses of SK-09 tablets in healthy adult participants.

Part 2 is a randomized, double-blind, placebo-controlled MAD study designed to evaluate the safety, tolerability, PK, and PD of multiple oral doses of SK-09 tablets in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 18 to 55 years (inclusive) at the time of screening.
2. Weight and BMI for female and male participants:

   Body weight ≥ 50 kg; Body mass index (BMI) between 18.5 and 29.9 kg/m2 (inclusive)
3. Participants must be in good general health.
4. Capable of understanding and voluntarily providing written informed consent prior to any study-related procedures.
5. Participants must have no plans for conception during the trial and for 3 months after the last dose, and must voluntarily use effective contraception with no plans for sperm or egg donation .

Exclusion Criteria:

1. History or current presence of clinically significant Cardiovascular; Respiratory ; Gastrointestinal; Neurological ; Hematologic/immunologic disorders.
2. Chronic GI conditions requiring daily medication; or history of bariatric surgery.
3. Live/attenuated vaccines within 4 weeks prior to dosing or planned during study.
4. Systolic blood pressure < 90 mmHg or ≥ 140 mmHg, or diastolic blood pressure ≥80 mmHg.
5. History of myocardial infarction, angina, coronary artery bypass grafting, angioplasty, stenting, congestive heart failure, uncontrolled hypotension, unexplained arrhythmia, ventricular tachycardia, atrioventricular block, QT prolongation syndrome, or symptoms/family history of QT prolongation syndrome, as assessed by the investigator to be unsuitable for participation.
6. Positive results for hepatitis B surface antigen, syphilis-specific antibodies, hepatitis C antibodies, or HIV antibodies.
7. Major surgery or trauma requiring hospitalization within 6 months.
8. Hypersensitivity to any component of SK-09 or its excipients.
9. Poor venous access or needle phobia impacting study procedures.
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months.
11. Current smokers unwilling to abstain during study.
12. Participants with ANY of the following abnormalities in clinical laboratory tests at screening and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥ 1.5×ULN;
    * Total bilirubin level ≥ 1.5×ULN (except Gilbert's with direct bilirubin ≤ ULN)
13. Blood loss or donation exceeding 400 mL within 3 months of dosing.
14. Other investigational product within 30 days of dosing or 5 half-lives (whichever longer).
15. Use of any medications, including over-the-counter drugs, herbal medicine, vitamins, and health supplements, within 2 weeks prior to the first dose or 5 half-lives (whichever longer).
16. Positive pregnancy test or breastfeeding.
17. Unprotected sexual activity within 2 weeks prior to the first dose.
18. Any condition that, in the investigator's opinion, may pose a safety risk to the participant, interfere with the study, or prevent the participant from completing the study or complying with its requirements (due to administrative or other reasons).
19. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation | up to 8 days post-dosing for SAD and up to 20 days post-dosing for MAD
  Number of participants with AE, with abnormal Vital Signs, abnormal Physical Examination findings, abnormal Laboratory Tests results, abnormal 12-lead ECG readings

SECONDARY OUTCOMES:
PK Evaluation（Cmax） | up to 72 hours post-dosing for SAD and up to 16 days post-dosing for MAD
  Pharmacokinetic characteristics after administration (Cmax）
PK Evaluation（Tmax） | up to 72 hours post-dosing for SAD and up to 16 days post-dosing for MAD
  Pharmacokinetic characteristics after administration
PK Evaluation（ AUC0-T） | up to 72 hours post-dosing for SAD and up to 16 days post-dosing for MAD
  Pharmacokinetic characteristics after administration (AUC0-T）
PK Evaluation ( AUC0-∞） | up to 72 hours post-dosing for SAD and up to 16 days post-dosing for MAD
  Pharmacokinetic characteristics after administration ( AUC0-∞）
PD evaluation | up to 12 hour post-dosing on Day 1 for SAD and pending for MAD
  urinary Rac1 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Ltd., Herston, Queensland, Australia